CLINICAL TRIAL: NCT01721642
Title: A Pilot Study to Evaluate the Safety and Efficacy of the Apica Access, Stabilization and Closure (ASC™) Device During and After Transcatheter Aortic Valve Implantation (TAVI) Procedures
Brief Title: A Pilot Study to Evaluate the Safety and Efficacy of the Apica Access, Stabilization and Closure (ASC™) Device
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Apica Cardiovascular Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-DP1
Record Dates: First submitted 2012-09-25; First posted 2012-11-06 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Aortic Valve Stenosis
Keywords: access; closure; trans-apical; trans-catheter aortic valve implantation; TAVI; trans-catheter aortic valve repair; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apica Cardiovascular ASC Device (Experimental): Access, stabilisation and closure with the Apica Cardiovascular ASC Device
  Interventions: Device: Apica Cardiovascular ASC Access, Stability and Closure Device

INTERVENTIONS:
Device: Apica Cardiovascular ASC Access, Stability and Closure Device — Access, stabilisation and closure of trans-apical approach for TAVI
  Other Names: Apica Cardiovascular, ASC

SUMMARY:
A pilot study to evaluate the safety and efficacy of the Apica Access, Stabilization, and Closure Device for accessing and closing the left ventricular apex during and after Transcatheter Aortic Valve Implantation (TAVI) procedures. Follow-up assessment will be made post-procedure, at 30 days and 90 days as well as longer term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥ 18 years of age.
* Subjects will be selected in accordance with the investigating centers standard operating procedures for TAVI subject selection and treatment. Subjects selected will meet all of the TAVI inclusion criteria as follows:

  * Subject has Senile degenerative aortic stenosis with echocardiography derived criteria: mean gradient > 40 mm Hg or jet velocity > 4.0 m/s or an aortic valve area (AVA) of < 0.8 cm2 (or AVA index < 0.5 cm2/m2.
  * Subject is symptomatic due to aortic valve stenosis as demonstrated by NYHA Functional Class > II.
  * Additive EuroScore > 9
  * Aortic annulus diameter > 21mm to < 27mm by TEE
  * The subject or the subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
  * The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.
  * The subject, after formal consults by a cardiologist and two cardiovascular surgeons agreed that medical factors precluding operation, based on a conclusion that the probability of death or serious, irreversible morbidity exceeded the probability of meaningful improvement. Specifically the probability of death or serious, irreversible morbidity exceeded 50%.

Exclusion Criteria:

Subjects will be selected in accordance with the investigating centers standard operating procedures for TAVI subject selection and treatment. The following TAVI exclusion criteria shall apply:

* Evidence of an acute myocardial infarction < 1 month before the intended treatment
* Aortic valve is a congenital unicuspid or bicuspid valve; or is non-calcified
* Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation > 3+)
* Pre-existing prosthetic heart valve in an position, prosthetic ring, or severe (greater than 3+) mitral insufficiency
* Blood dyscrasias as defined: Leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy.
* Untreated clinically significant coronary artery disease requiring revascularization
* Hemodynamic instability requiring inotropic therapy or mechanical hemodynamic support devices
* Need for emergency surgery for any reason
* Hypertrophic cardiomyopathy with or without obstruction
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Active peptic ulcer or upper gastro-intestinal bleeding within the prior 3 months
* A known hypersensitivity of contraindication to asprin, heparin, ticlopidine (Ticlid), or clopidogrel (Plavix), or sensitivity to contrast media, which cannot be adequately pre-medicated
* Recent (within 6 months) cerebrovascular accident or transient ischemic attack
* Renal insufficiency and/or end stage renal disease requiring chronic dialysis.
* Life expectancy < 12 months due to non-cardiac co-morbid conditions.

The following ASC device exclusion criteria shall apply:

* Subjects with <10mm Left ventricular wall thickness at apical access site
* LVEF < 30%
* Subject with previous DOR procedure
* Subject access site has less than 2 cm squared "fat" free area under visual observation
* Subject has known Allergy or hypersensitivity to Titanium
* Subject requires MR Imaging post procedure
* Subject is Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Access safety | Within 2 hours from initial skin incision
  Observation of no myocardial tearing on entry of the device
Closure safety | Within 2 hours from initial skin incision
  Observation of no acute post-procedural bleeding or pericardial effusion.

SECONDARY OUTCOMES:
Investigational device performance: LV function | 24 hours, 30 days and 90 days post-procedure
  % LVEF no worse than baseline as assessed by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walther, Prof, Principal Investigator — Kerckhoff Klinik